CLINICAL TRIAL: NCT00910143
Title: Introduction of Total Mesorectal Excision (TME) in the Treatment of Rectal Cancer. Influence of This New Operation Technique on Local Recurrence and Long-Time Survival. Retrospective Study: 1993-2001
Brief Title: Introduction and Influence of Total Mesorectal Excision (TME) in the Treatment of Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Pietro Renzulli MD, Bern University Hospital, Departement of visceral Surgery
Other Study IDs: KEK 08-05-09
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Colorectal Surgery; Surgery; Local neoplasm recurrence; survival; Follow-up Study
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients operated before summer 1995, that is before the introduction of TME
  Interventions: Procedure: conventional rectal surgery
- 2: patients operated after summer 1995, that is after the introduction of TME.
  Interventions: Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: conventional rectal surgery — type of rectal surgery before the introduction of TME
  Groups: 1
Procedure: total mesorectal excision — total mesorectal excision
  Groups: 2

SUMMARY:
Total mesorectal excision (TME) is a rather new operation technique in the treatment of rectal cancer. It is known to reduce the rate of local recurrences. However, the influence on long-term survival is unclear.

DETAILED DESCRIPTION:
Background

The TME technique for rectal cancer surgery was introduced in our department in summer 1995. TME is known to reduce the rate of local recurrences. However, its influence on long-term survival in unclear.

All patients with rectal cancer from 1993 to 2001 are reviewed. The patients charts are reviewed and the following main characteristics are retrieved: age, gender, time of operation, operation technique, tumor stage, tumor localisation, tumor size, neoadjuvant or adjuvant treatment, complications, follow-up with respect to the appearance of local recurrences and distant metastases.

Comparison of two groups of patients. Group 1: patients operated before summer 1995, that is before the introduction of TME. Group 2: patients operated after summer 1995, that is after the introduction of TME.

Objective

Study the influence of a new operation method (TME) on outcome (local recurrence, survival).

Methods

All patients with rectal cancer from 1993 to 2001 are reviewed. The patients charts are reviewed and the following main characteristics are retrieved: age, gender, time of operation, operation technique, tumor stage, tumor localisation, tumor size, neoadjuvant or adjuvant treatment, complications, follow-up with respect to the appearance of local recurrences and distant metastases.

Comparison of two groups of patients. Group 1: patients operated before summer 1995, that is before the introduction of TME. Group 2: patients operated after summer 1995, that is after the introduction of TME.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the rectum
* 16 years and older

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all adult patients with adenocarcinoma of the rectum who underwent colorectal surgery at Bern University Hospital between January 1993 and December 2001
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 1993-01; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Local recurrence, recurrence-free survival, overall survival | 6 months and 1, 2, 3, 4 and 5 years after the operation

SECONDARY OUTCOMES:
Surgical complications | first 30 days after the operation
quality of life
Percentage of patients undergoing transcatheter arterial embolisation

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Renzulli, MD, Principal Investigator — Bern University Hospital, 3010 Bern, Switzerland
Locations (1):
- Dep. of visceral and transplant surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Heald RJ. Total mesorectal excision is optimal surgery for rectal cancer: a Scandinavian consensus. Br J Surg. 1995 Oct;82(10):1297-9. doi: 10.1002/bjs.1800821002. No abstract available. PMID 7489148
- [Background] Mella J, Biffin A, Radcliffe AG, Stamatakis JD, Steele RJ. Population-based audit of colorectal cancer management in two UK health regions. Colorectal Cancer Working Group, Royal College of Surgeons of England Clinical Epidemiology and Audit Unit. Br J Surg. 1997 Dec;84(12):1731-6. PMID 9448628
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] Maurer CA, Renzulli P, Meyer JD, Buchler MW. [Rectal carcinoma. Optimizing therapy by partial or total mesorectum removal]. Zentralbl Chir. 1999;124(5):428-35. German. PMID 10420530
- [Background] Heald RJ, Moran BJ, Ryall RD, Sexton R, MacFarlane JK. Rectal cancer: the Basingstoke experience of total mesorectal excision, 1978-1997. Arch Surg. 1998 Aug;133(8):894-9. doi: 10.1001/archsurg.133.8.894. PMID 9711965
- [Background] Laurent C, Nobili S, Rullier A, Vendrely V, Saric J, Rullier E. Efforts to improve local control in rectal cancer compromise survival by the potential morbidity of optimal mesorectal excision. J Am Coll Surg. 2006 Nov;203(5):684-91. doi: 10.1016/j.jamcollsurg.2006.07.021. Epub 2006 Sep 20. PMID 17084330
- [Background] Kapiteijn E, Putter H, van de Velde CJ; Cooperative investigators of the Dutch ColoRectal Cancer Group. Impact of the introduction and training of total mesorectal excision on recurrence and survival in rectal cancer in The Netherlands. Br J Surg. 2002 Sep;89(9):1142-9. doi: 10.1046/j.1365-2168.2002.02196.x. PMID 12190680
- [Background] Bernardshaw SV, Ovrebo K, Eide GE, Skarstein A, Rokke O. Treatment of rectal cancer: reduction of local recurrence after the introduction of TME - experience from one University Hospital. Dig Surg. 2006;23(1-2):51-9. doi: 10.1159/000093494. Epub 2006 May 23. PMID 16717469